CLINICAL TRIAL: NCT05216848
Title: Prevalence and Risk Factors for Serious Birth Concerns in Unselected Population of Mothers
Acronym: RiskfSBC
Status: Completed | Type: Observational
Sponsor: Comenius University (Other)
Responsible Party: Sponsor
Other Study IDs: EC/188/2021/UNBRuzinov
Record Dates: First submitted 2022-01-19; First posted 2022-02-01 (Actual); Last update posted 2023-05-01 (Actual); Status verified 2023-04

CONDITIONS: Serious Concerns
Keywords: fear of childbirth; Wijma Delivery Expectancy Questionnaire

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- nulliparas with no existing complications in the third trimester: The investigators involve every nullipara giving birth in a period of two years.
  Exclusion criteria: unwilling to participate, minors (under 18 years old), high risk pregnancy, foetus mortus or perinatal death of the newborn, with slovak language
  Interventions: Other: Wijma Delivery Expectancy Questionnaire; Other: Clinical data collection
- multiparas with no existing complications in the third trimester: The investigators involve every multipara giving birth in a period of two years.
  Exclusion criteria: unwilling to participate, minors (under 18 years old), high risk pregnancy, foetus mortus or perinatal death of the newborn, with slovak language, previous caesarean section
  Interventions: Other: Wijma Delivery Expectancy Questionnaire; Other: Clinical data collection

INTERVENTIONS:
Other: Wijma Delivery Expectancy Questionnaire — Simple questionaire identifying the level of fear of childbirth in pregnancy
Other: Clinical data collection — Collection of the standard clinical data during hospitalization

SUMMARY:
The aim of this study is to determine the prevalence of significant concerns about childbirth and their impact on the course and outcome of childbirth. By identifying a group of mothers who have an excessive fear of childbirth, the occurrence of surgical births can be influenced by the right intervention.

DETAILED DESCRIPTION:
The fear of childbirth is one of the most common mental health concerns during pregnancy. Elevated levels of anxiety during childbirth may lead to increased risk of elective caesarean section or prolonged labour. About 80% of pregnant women suffer from certain kind of childbirth fear. The most commonly used tool for assessment and diagnosis of childbirth fear is Wijma Delivery Expectance Questionnaire (WDEQ). This questionnaire has been translated and validated into several languages. In 2020 the Slovak version of the questionnaire was validated. All women who completed antenatal counseling at 36 weeks of gestation were included in the cohort. A slovak version of questionnaire was issued to all women and the results were recorded in the protocol. Subsequently, demographic data, medical facts and childbirth outcome were added from the medical documentation. The results of the birth were compared with the results of the questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* The investigators involve every nullipara and multipara giving birth at 2nd Department of Obstetrics and Gynecology, University Hospital Bratislava and Comenius University, Bratislava, Slovak Republic in a period of two years

Exclusion Criteria:

* unwilling to participate, minors (under 18 years old), high risk pregnancy, foetus mortus or perinatal death of the newborn, with slovak language, previous Caesarean section (for multipara)

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — primipara giving birth
Study Population: Total 700 nullipara and multipara giving birth at 2nd Department of Obstetrics and Gynecology, University Hospital Bratislava and Comenius University, Bratislava, Slovak Republic in a period of two years
Sampling Method: Non-Probability Sample
Enrollment: 700 (Actual)
Dates: Start 2019-09-01 (Actual); Primary Completion 2022-12-01 (Actual); Study Completion 2023-03-30 (Actual)

PRIMARY OUTCOMES:
Significant fear of childbirth | 15 minutes
  Identifying the level of fear of childbirth in pregnancy by using a most widely used tool Wijma Delivery Expectancy Questionnaire

CONTACTS AND LOCATIONS:
Locations (1):
- 2nd Department of Obstetrics and Gynecology, University Hospital Bratislava and Comenius University, Bratislava, Slovak Republic, Bratislava, Slovak Republic, Slovakia

IPD SHARING:
Plan to Share IPD: No